CLINICAL TRIAL: NCT00493233
Title: Antipsychotic Polypharmacy in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Psychiatric Research Foundation (Other)
Responsible Party: Dr. David Mamo, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 174/2006
Record Dates: First submitted 2007-06-04; First posted 2007-06-28 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia; antipsychotics; polypharmacy; double-blind; randomized
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Clozapine; Quetiapine Fumarate; Haloperidol; Perphenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: 2 antipsychotic medications (combinations of olanzapine, risperidone, clozapine, seroquel, haldol, perphenazine)
- 2 (Placebo Comparator)
  Interventions: Drug: main antipsychotic medication and placebo

INTERVENTIONS:
Drug: 2 antipsychotic medications (combinations of olanzapine, risperidone, clozapine, seroquel, haldol, perphenazine) — Primary antipsychotic medication (olanzapine, oral risperidone, seroquel, clozapine, haldol, perphenazine) will be determined by the treating physician and participants will continue taking the concomitant antipsychotic drug. The dose of the main antipsychotic drug will remain open and flexible at the discretion of the attending physician. The dose of the "second" antipsychotic drug will remain fixed throughout the study period.
  Arms: 1
Drug: main antipsychotic medication and placebo — The "main" antipsychotic drug will be determined by the treating physician. Participants will be allocated to placebo in place of the concomitant antipsychotic drug. The dose of the "main" antipsychotic drug will remain open and flexible at the discretion of the attending physician.
  Arms: 2

SUMMARY:
The literature suggests that when a patient is prescribed more than one antipsychotic for at least 30 days, he or she is likely to continue on that combination. In this 12 week study 100 adult patients being treated on more than one antipsychotic medication for at least 30 days will be recruited. In order to control for the natural course of the illness, patients will be randomly assigned to one of two groups: the first group will continue the second medication hidden in a capsule at the same dose, while the second group will be given an inactive capsule (placebo) - the capsules in both group will be identical such that neither the patient nor the treating doctor will be able to identify the group assignment.

DETAILED DESCRIPTION:
There is no evidence that using more than one antipsychotic drug enhances clinical efficacy. Nonetheless, this practice is highly prevalent (up to 1/3 of our patient population), and physicians are reluctant to reduce patients' treatment to a single antipsychotic drug for fear of precipitating relapse. This study therefore seeks to evaluate the effectiveness of continued treatment with more than one antipsychotic drug using a rigorous placebo-controlled design. The results of this study will subsequently serve to guide physicians in making appropriately informed decisions regarding the continuation of multiple antipsychotic drugs.

Our primary hypothesis is that we expect to find no difference in the primary variable of interest (BPRS) following reduction to antipsychotic monotherapy (placebo group) versus continuing antipsychotic polypharmacy.

This proposed study is the first study to systematically address the reduction of antipsychotic polypharmacy to monotherapy in patients with primary psychotic disorders in a prospective, double-blind, placebo-controlled design. The results of this study will have important implications for the clinical practice of physicians treating the severely mentally ill who are often constrained to practice beyond the limits of available clinical guidelines and evidence based medicine. Thus, in light of the high and growing prevalence of this practice, the proposed study speaks to a real and practical clinical dilemma within this field. Furthermore, as a university-based, tertiary care psychiatric centre serving thousands of severely ill patients suffering from primary psychotic disorders and with an established track record for innovative clinical research, we are uniquely placed to address these critical questions.

Male or female subjects aged ≥ 18 years suffering from a primary psychotic disorder treated with two antipsychotic drugs for at least 30 days (excluding "prn" or "as needed" antipsychotic prescriptions) will be eligible to participate in this study. Subjects with a history of treatment with a depot antipsychotic within 6-months of enrollment will be excluded form the study unless the depot antipsychotic is considered the "main" antipsychotic drug in this study. The "main" antipsychotic drug will be determined by the treating physician, except for the case of clozapine which will be considered the 'main' antipsychotic. Eligible subjects will be randomly allocated to two groups: Group 1 will continue taking the concomitant antipsychotic drug; Group 2 will be allocated to placebo in place of the concomitant antipsychotic drug. The dose of the "main" antipsychotic drug will remain open and flexible at the discretion of the attending physician. The dose of the "second" antipsychotic drug will remain fixed throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years
* Suffering from a primary psychotic disorder (confirmed using the MINI International Neuropsychiatric Interview for DSM-IV (Version 5.0.0)
* Treated with two antipsychotic drugs for at least 30 days (excluding "prn" or "as needed" antipsychotic prescriptions)

Exclusion Criteria:

* A history of treatment with a depot antipsychotic within 6-months of enrollment will be excluded form the study unless the depot antipsychotic is considered the "main" antipsychotic drug in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | intermittent
Clinical Global Impression Scale | intermittent

SECONDARY OUTCOMES:
Barned Akathisia Scale | intermittent
Simpson-Angus Scale (SAS) | intermittent

CONTACTS AND LOCATIONS:
Overall Officials: David Mamo, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Borlido C, Remington G, Graff-Guerrero A, Arenovich T, Hazra M, Wong A, Daskalakis ZJ, Mamo DC. Switching from 2 antipsychotics to 1 antipsychotic in schizophrenia: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2016 Jan;77(1):e14-20. doi: 10.4088/JCP.14m09321. PMID 26845273
- See also: Information about research at the Centre for Addiction and Mental Health (CAMH) — http://www.camh.net/research